CLINICAL TRIAL: NCT03166319
Title: The Utility of Intracranial Vessel Wall Imaging for Suspected CNS Vasculitis Diagnosis and Assessment of Disease Activity.
Brief Title: Vessel Wall Imaging for Diagnosis and Monitoring of Central Nervous System (CNS) Vasculitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vance Lehman, Assistant Professor of Radiology, Mayo Clinic, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-009297
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Vasculitis, CNS; Vasculitis, Cerebral
MeSH Terms: conditions — Vasculitis, Central Nervous System | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Patients with suspected primary CNS vasculitis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspected CNS Vasculitis (Experimental): Patients with suspected CNS vasculitis will undergo an MRI, including intracranial vessel wall imaging.
  Interventions: Diagnostic Test: MRI, including intracranial vessel wall imaging

INTERVENTIONS:
Diagnostic Test: MRI, including intracranial vessel wall imaging — MRI/MRA/intracranial high-resolution vessel wall imaging (HR-VWI)

SUMMARY:
This is a prospective pilot study to determine the utility of MRI and high resolution intracranial vessel wall imaging for the diagnosis and disease activity assessment of intracranial vasculitis.

DETAILED DESCRIPTION:
This study will evaluate patients with suspected primary angiitis of the central nervous system (PACNS), recruited during initial work-up by our multi-disciplinary team. Given the low incidence of CNS vasculitis and the fact that some patients are routed to a quaternary care center after initial work-up and diagnosis, evaluation of both groups will be useful to maximize the number of participants evaluated and to provide a representative sample of patients typically treated. During the study, participants will ultimately be deemed to have;

1. A specific clinical and pathologic subtype of PACNS,
2. PACNS not otherwise specified (NOS) without pathologic or clinical proof of a specific subtype, or
3. An alternative diagnosis other than PACNS.

Patients will undergo a standardized imaging and clinical examination at presentation and at pre-defined follow-up periods. Imaging examinations will include an MRI of the head, standard magnetic resonance angiogram (MRA) of the head, and intracranial vessel wall imaging without and with IV gadolinium. Patients will receive up to 4 imaging examinations at predefined intervals as part of this study. MRI/MRA/Vessel wall features will be evaluated by 2 neuroradiologists. Imaging findings will be correlated to clinical and any available laboratory or pathologic data. The target accrual is 10 patients for this pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is determined to have suspected PACNS upon evaluation by a neurologist or rheumatologist or may have an established diagnosis of PACNS of any duration as determined by a neurologist or rheumatologist.
2. Ability to undergo routine clinical testing, including lumbar puncture performed for PACNS to exclude potential alternative diagnoses (for initial suspected cases).
3. Ability to provide informed consent.

Exclusion Criteria:

1. Less than 18 years of age.
2. Any absolute contraindication to 3 Tesla MRI.
3. Any absolute contraindication to gadolinium.
4. Contraindication to lumbar puncture such as severe coagulopathy.
5. High risk carotid atherosclerotic plaque defined as either greater than 70% stenosis or known high risk plaque features such as intra-plaque hemorrhage.
6. Medium or high risk factors for cardioembolic stroke based on the Trial of Org 10172 in Acute Stroke Treatment (TOAST) criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Diagnosis of Stroke | Approximately 5 months after baseline
  Clinical or MRI evidence of stroke on follow-up exam.

CONTACTS AND LOCATIONS:
Overall Officials: Vance Lehman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials